CLINICAL TRIAL: NCT01712165
Title: Micronutrient-supplemented Milk Study in Women of Childbearing Age
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fonterra Research Centre (Industry)
Collaborators: Changi General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: FON-ALTHEA-SG-2012-01
Record Dates: First submitted 2012-10-19; First posted 2012-10-23 (Estimated); Last update posted 2013-10-11 (Estimated); Status verified 2013-10

CONDITIONS: Increase the Concentration of Folic Acid in Women of Childbearing Age
Keywords: Folic acid supplement; Neural tube defect-affected pregnancy; Homocysteine concentration; Plasma Folate concentration; Plasma vitamin B12 concentration

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- ANMUM Materna (Active Comparator): 75g milk powder in 400 ml water daily for 12 weeks.
  Interventions: Dietary Supplement: ANMUM Materna
- Control (Placebo Comparator): 75g of milk powder in 400 ml water for 12 weeks.
  Interventions: Dietary Supplement: Control (milk powder)

INTERVENTIONS:
Dietary Supplement: ANMUM Materna
  Arms: ANMUM Materna
Dietary Supplement: Control (milk powder)
  Arms: Control

SUMMARY:
The purpose of this study is to determine if consuming ANMUM Materna (a fortified milk product) over a 12-week period increases red blood cell folate concentrations in women of childbearing age in Singapore, compared to an equivalent amount of standard (unfortified) milk.

DETAILED DESCRIPTION:
Folic acid (~400 µg/day) taken around the time of conception significantly reduces the risk of a neural tube defect (NTD)-affected pregnancy. Strategies to reduce NTD with folic acid, include supplement use and food fortification. An attractive strategy for NTD prevention is the use of fortified foods targeted for use by women planning a pregnancy. Fonterra currently markets a fortified-milk (ANMUM Materna) in Asia, designed for use prior to and during pregnancy. This milk product, if consumed as directed, provides ~400 µg folic acid per day. It is not known whether ANMUM Materna will reduce NTD rate. However, in a case-control study the risk of NTD was inversely associated with maternal red blood cell (RBC) folate concentrations. Accordingly, if ANMUM Materna increases RBC folate, it could be expected to decrease NTD risk.

In this study, the ANMUM Materna fortified milk will be tested against a standard control (unfortified) milk over a 12 week period. The subjects will consume 75g of milk powder daily throughout the supplementation period.

ELIGIBILITY:
Inclusion Criteria:

* Female 21-35 years old.
* Able to understand the nature and purpose of the study, including potential risks and side effects.
* Willing to consent to study participation and to comply with study requirements.
* Negative Pregnancy test at screening

Exclusion Criteria:

* Consumption of vitamins and/or mineral supplements known to contain folate 6 months prior.
* Chronic disease.
* Milk and/or lactose-intolerant.
* Pregnancy in the last 12 months, or currently planning a pregnancy.
* Prior history of NTD-affected pregnancy
* Serum Folate deficiency

Ages: 21 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2013-06; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Increase in red blood cell folate concentration | 12 weeks
  To determine if consuming ANMUM Materna over a 12-week period increases red blood cell folate concentrations in women of childbearing age in Singapore, compared to an equivalent amount of standard (unfortified) milk.

SECONDARY OUTCOMES:
Reduction in homocysteine concentration | 12 weeks
  To determine if consuming ANMUM Materna over a 12-week period lowers homocysteine concentrations in women of childbearing age, compared to an equivalent amount of standard (unfortified) milk.
Increase in plasma folate concentration | 12 weeks
  To determine if consuming ANMUM Materna over a 12-week period increases plasma folate concentrations in women of childbearing age, compared to an equivalent amount of standard (unfortified) milk.
Increase in plasma vitamin B12 concentration | 12 weeks
  To determine if consuming ANMUM over a 12-week period increases plasma vitamin B12 concentrations in women of childbearing age, compared to an equivalent amount of standard (unfortified) milk.

CONTACTS AND LOCATIONS:
Overall Officials: Magdalin Cheong, Principal Investigator — Changi General Hospital
Locations (1):
- Changi General Hospital, Singapore, Singapore